CLINICAL TRIAL: NCT06840158
Title: A Double-blind Comparative Randomized Trial to Evaluate the Safety and Efficacy of the Drug Miotox® in Children with Cerebral Palsy
Brief Title: Double-blind Comparative Randomized Multicenter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: № MTK-III-D-DCP-04/2019
Record Dates: First submitted 2025-01-27; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy (CP)
Keywords: botulinum toxin
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Miotox®(Botulinum toxin type A is a hemagglutinin complex) (Experimental): Children of the younger age group from 2 to 12 years (2 years 0 months 0 days - 11 years 11 months 29 days) Group 1 - 40 children who were injected with the drug Miotox®;
  Interventions: Drug: Miotox (Botulinum toxin type A is a hemagglutinin complex)
- Botox (Botulinum toxin type A - hemagglutinin complex - 100 units) (Active Comparator): Children of the younger age group from 2 to 12 years (2 years 0 months 0 days - 11 years 11 months 29 days) Group 2 - 40 children who were injected with Botox®.
  Interventions: Drug: BOTOX®

INTERVENTIONS:
Drug: Miotox (Botulinum toxin type A is a hemagglutinin complex) — During the study, patients were injected with the investigational drug Miotox® .
  For the treatment of spasticity and equine varus deformity of the foot in children with cerebral palsy, drugs were injected into two points of each head of the calf muscle (medial and lateral). In case of damage to one limb, the total dose was 4 units / kg of body weight per affected limb. In diplegia, the total dose was 6 units / kg of body weight for both affected limbs. The total total dose should not exceed 200 units.
  This course of treatment is based on the current instructions for the medical use of Botox®.
  Arms: Miotox®(Botulinum toxin type A is a hemagglutinin complex)
Drug: BOTOX® — During the study, patients were injected with the investigational comparison drug Botox®.
  For the treatment of spasticity and equine varus deformity of the foot in children with cerebral palsy, drugs were injected into two points of each head of the calf muscle (medial and lateral). In case of damage to one limb, the total dose was 4 units / kg of body weight per affected limb. In diplegia, the total dose was 6 units / kg of body weight for both affected limbs. The total total dose should not exceed 200 units.
  This course of treatment is based on the current instructions for the medical use of Botox®.
  Arms: Botox (Botulinum toxin type A - hemagglutinin complex - 100 units)

SUMMARY:
The name of the study: is a double-blind comparative randomized trial to evaluate the safety and efficacy of the drug Miotox® with the participation of children with cerebral palsy The code/number of the Protocol No. MTK-III-D-cerebral palsy-04/2019, version 5.0 dated 09/01/2021.

Investigational drug Trade Name: Miotox®. Description: Transparent or slightly opalescent liquid from colorless to light yellow. Manufacturer: FSBI "M.P. Chumakov FNCRIP RAS", Russia Comparison drug: Trade Name: Botox® Description: dried white substance in the form of a barely noticeable film located at the bottom of the bottle. Manufacturer: Allergan Pharmaceuticals Ireland, Ireland.

The studied indication for use is Focal spasticity associated with dynamic foot deformity of the "horse foot" type due to spasticity in patients 2 years and older with cerebral palsy who are on outpatient treatment Study design Double-blind comparative randomized multicenter The sponsor of the study is Innopharm LLC, Russia Clinical Development: Phase III The start date of the study is 10/15/2021. The date of completion of the study is 06/29/2022.

ELIGIBILITY:
Inclusion Criteria:

All patients were checked for compliance with the following inclusion criteria:

* Written and dated Informed consent of the child's parent to participate in the clinical trial; The age of the child is from 2 to 12 years (2 years 0 months 0 days - 11 years 11 months 29 days);
* Focal spasticity associated with dynamic foot deformity of the "horse foot" type due to spasticity in children with cerebral palsy undergoing outpatient treatment;
* The degree of spasticity on the modified Ashworth scale (MAS) 2 or more;
* Grade level on the scale of basic motor functions for cerebral palsy, extended and refined version (GMFCS - E&R) I - III;
* Children and their parents who are able to fulfill the requirements of the Protocol (i.e., fill out a self-observation diary, come to control visits).

Exclusion Criteria:

During the study, patients were excluded if any of the following criteria were present:

* Withdrawal of Informed consent by the patient's parent;
* Serious adverse events or adverse events that do not meet the criteria of severity, in the development of which, in the opinion of the researcher, further participation in the study may be detrimental to the health or well-being of the patient;
* The need for procedures and/or drug treatment that are not permitted by the Protocol of this study;
* The patient was included in violation of the criteria for inclusion/non-inclusion of the Protocol;
* The appearance of non-inclusion criteria during the study;
* The need for surgical intervention.
* The patient's incompetence with the examination procedures.
* Any condition of the patient that requires, in the reasonable opinion of the research physician, the withdrawal of the patient from the study;
* The patient refuses to cooperate or is undisciplined (for example, the patient does not show up for a scheduled visit without warning the researcher and/or loss of communication with the patient);
* The patient is out of observation;
* Non-compliance by the patient with the established Protocol requirements, rules of stay at the clinical base; For administrative reasons (termination of the study by the Sponsor or regulatory authorities), as well as in case of gross violations of the Protocol that may affect the results of the study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Safety assessment | 14 weeks
  The frequency of adverse events during the study:
  adverse events of an immediate type (allergic reactions) that occur within 2 hours after administration of the drug under study and identified both by the researcher and according to information provided to the researcher by the patient's parent; adverse events (local and systemic reactions) that occur within 7 days after administration of the test drug and are identified according to information provided to the researcher by the patient's parent; other adverse events that occur 7 days after administration of the test drug (from 8 to 84 days after administration of the test drug, without taking into account the permissible interval of visits) and noted by the patient's parent in the Self-observation Diary.
Efficasy assessment | 14 weeks
  The change in the level of spasticity (decrease in score) on the Modified Ashworth Scale (MAS) scale at week 4 compared to the baseline level from 1 to 4 points.

SECONDARY OUTCOMES:
Safety assessment | 14 weeks
  The frequency of serious adverse events during the study.
Safety assessment | 14 weeks
  The frequency of adverse events and serious adverse events, at least probably related to the study drug during the study.
Safety assessment | 14 weeks
  Cases of early termination of patients' participation in the study due to the development of NYA/NYA associated with the use of research drugs.
Efficasy assessment | 14 weeks
  Change in the level of spasticity on the Modified Ashworth Scale (MAS) scale (decrease in score) at 1, 8 and 12 weeks compared to the baseline level.
Efficasy assessment | 14 weeks
  Severity of pain on a 10-point Visual Analogue Scale (VAS) at 1, 4, 8 and 12 weeks compared to the baseline level (decrease in pain severity).
Efficasy assessment | 14 weeks
  The state of motor functions according to the scale of basic motor functions for cerebral palsy (GMFCS - E&R) at 1, 4, 8 and 12 weeks compared with the baseline level.
Efficasy assessment | 14 weeks
  Measurement of spasticity on the Mental Toughness Scale (MTS )(decrease in score) at 1, 4, 8 and 12 weeks compared to the baseline level.

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - SPb GBUZ "DGP No. 45 of the Nevsky district, Saint Petersburg
  - GBUZ SODKB named after N.N. Ivanova, Candidate of Medical Sciences;, Samara
  - Limited Liability Company "Santerra" (LLC "Santerra"), Stavropol